CLINICAL TRIAL: NCT03144284
Title: Assessment of Knowledge, Attitude, and Practice of Minimal Intervention Dentistry in a Group of Dental Interns in Egypt: A Cross-sectional Study
Brief Title: Assessment of Knowledge, Attitude, and Practice of Minimal Intervention Dentistry in a Group of Dental Interns
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Hassan Hashim, Principal Investigator, pediatric dentistry master degree student, Cairo University
Other Study IDs: Noha Hasan Mohamed Hashim
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental interns: dental interns in pediatric dentistry department, faculty of dentistry, Cairo University.
  Interventions: Other: Knowledge, attitude, and practice survey

INTERVENTIONS:
Other: Knowledge, attitude, and practice survey — A knowledge, attitude, and practice questionnaire is going to be distributed to dental interns.
  Other Names: KAP survey

SUMMARY:
Minimal intervention dentistry (MID) is a modern medical approach that aims to maximize preservation of healthy dental tissues. When operative intervention is required it is as minimally invasive as possible. This study will assess the knowledge of a group of dental interns regarding minimal intervention dentistry in Egypt and whether this knowledge is translated into positive attitude and practice among them.

DETAILED DESCRIPTION:
Healthy oral tissues enable the child to eat, speak and socialize which contributes to general wellbeing. Dental caries during childhood is a major public health problem and throughout the 20th century, the dominant practice patterns of managing dental caries relied on the purely surgical approach of G.V Black such as the concept of "extension for prevention". One of the drawbacks of this approach is an unnecessary removal of healthy oral tissues.

Comprehensive knowledge of dental cariology, advances in dental restorative materials and modern diagnostic devices are changing pediatric restorative dentistry.

minimal intervention dentistry (MID) is a modern medical approach that aims to maximize preservation of healthy dental tissues based on individualized patient care of early detection of disease, risk assessment diagnosis, and prevention. When operative intervention is required it is as minimally invasive as possible.

There is insufficient information about knowledge and practice of modern dental approaches including minimal intervention dentistry among dental interns in Egypt. Available studies concerned with this subject were not done in Egypt.

Due to this shortage of information, the application of MID in the Egyptian society cannot be fully assessed, and problems associated with its practice cannot be identified and solved. This shortage of information may also deprive children of getting benefits of MID.

Thus; this study will assess the knowledge of a group of dental interns regarding minimal intervention dentistry in Egypt, and whether this knowledge is translated into positive attitude and practice among them.

Knowledge, attitude, and practice (KAP) surveys can be used to identify knowledge gaps and culturally related misconceptions of new health approaches or interventions. They can determine factors influencing behaviors that are not known, and how and why people practice certain health behaviors.

KAP surveys can be also used to identify needs, problems and barriers, as well as solutions for improving quality and accessibility of health services by studying factors and possible determinants influencing treatment decisions.

This study aims to identify deficiencies (if present) in knowledge, attitude, and practice of MID among a group of dental interns in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Dental interns attending pediatric dentistry in the faculty of dentistry, Cairo University.

Exclusion Criteria:

* Interns refusing to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dental interns are fresh dental graduates who must attend an official clinical training before getting a licence to practice dentistry.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practice mean score | Through study completion, an average of 1 year.
  Scores will be calculated according to the options selected by dental interns. The primary outcome is the mean score of the knowledge, attitude and practice survey.

SECONDARY OUTCOMES:
response rate | Through study completion, an average of 1 year.
  percentage of dental interns who agree to participate in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Noha Hasan Mohamed Hashim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are not going to be shared. The names of dental interns are going to be replaced by codes during data collection.

REFERENCES:
- [Result] Gaskin EB, Levy S, Guzman-Armstrong S, Dawson D, Chalmers J. Knowledge, attitudes, and behaviors of federal service and civilian dentists concerning minimal intervention dentistry. Mil Med. 2010 Feb;175(2):115-21. doi: 10.7205/milmed-d-09-00140. PMID 20180481
- [Result] Leal SC. Minimal intervention dentistry in the management of the paediatric patient. Br Dent J. 2014 Jun 13;216(11):623-7. doi: 10.1038/sj.bdj.2014.449. PMID 24923936